CLINICAL TRIAL: NCT05323214
Title: Comparative Study Between Dexmedetomidine and Fentanyl as Adjuvants to Bupivacaine for Post-operative Epidural Analgesia in Abdominal Surgeries
Brief Title: Comparative Study Between Two Adjuvant Drugs to Bupivacaine for Post-operative Epidural Analgesia in Abdominal Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU MD 121/2021
Record Dates: First submitted 2022-01-21; First posted 2022-04-12 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Epidural Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Normal saline 2 ml will be mixed with 48 ml bupivacaine 0.125% in an elastomeric pump. The rate of epidural infusion will be 5ml/hr for the postoperative 24 hours.
  Interventions: Drug: Control Analgesic regimen
- Fentanyl group (Other): Fentanyl 2 ml (100 μg) will be mixed with 48 ml bupivacaine 0.125% in an elastomeric pump. The rate of epidural infusion will be 5ml/hr for the postoperative 24 hours.
  Interventions: Drug: Fentanyl Analgesic regimen
- Dexmedetomidine group (Other): Dexmedetomidine 1 ml (100 μg) plus 1 ml normal saline will be mixed with 48 ml bupivacaine 0.125% in an elastomeric pump. The rate of epidural infusion will be 5ml/hr for the postoperative 24 hours.
  Interventions: Drug: Dexmedetomidine Analgesic regimen

INTERVENTIONS:
Drug: Control Analgesic regimen — testing the efficiency of bupivacaine without adjuvant drugs in epidural analgesia
  Other Names: Epidural Bupivacaine
  Arms: Control group
Drug: Fentanyl Analgesic regimen — testing the efficiency of Fentanyl as an adjuvant drug to bupivacaine in epidural analgesia
  Other Names: Epidural Fentanyl Bupivacaine
  Arms: Fentanyl group
Drug: Dexmedetomidine Analgesic regimen — testing the efficiency of Dexmedetomidine as an adjuvant drug to bupivacaine in epidural analgesia
  Other Names: Epidural Dexmedetomidine Bupivacaine
  Arms: Dexmedetomidine group

SUMMARY:
Epidural analgesia is associated with early postoperative mobilization and rehabilitation with minimally associated pain and discomfort. Analgesic effect of local anesthetics is augmented by addition of adjuvants in epidural anesthesia ensuring satisfactory postoperative period. This study evaluates the effect of dexmedetomidine and fentanyl as additives to bupivacaine for epidural analgesia.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of dexmedetomidin and fentanyl as adjuvants to bupivacaine for postoperative epidural analgesia in abdominal surgeries regarding block characteristics, post-operative analgesia, hemodynamic changes and any anticipated side effects.

* Type of Study: Prospective randomized comparative clinical study.
* Study Setting: The operating theatres of Ain Shams University Hospitals
* Study Period: One year
* Sampling Method: Random sampling Patients randomly allocated by computer generated randomization and using opaque sealed envelopes to one of the three study groups according to the adjuvant drug used in postoperative analgesia.
* Sample Size: Total 75 cases divided into 25 cases in each group. Kiran et al. (2018) reported a rather large effect size comparing onset to sensory block and time to maximum motor block. In a one-way ANOVA study, sample sizes of 25 cases per group in three groups whose means are to be compared. The total sample of 75 subjects achieves 80% power to detect differences among the means versus the alternative of equal means using an F test with a 0.0500 significance level. The size of the variation in the means is represented by the effect size = 0.4

ELIGIBILITY:
Inclusion Criteria:

* ASA I or ASA II patients.
* Age group: 21-70 years old.
* BMI ≤40
* Duration of procedure ≤ 180 minutes.

Exclusion Criteria:

* Patients with known neurologic and psychiatric illness will be excluded from the study.
* Contraindications for epidural anesthesia as patient refusal, bleeding or coagulation test abnormalities, local skin infection at spinal lumbar region, raised intracranial pressure and hypovolemia
* Spine abnormalities.
* Systemic disorders like hematological, respiratory, cardiac, renal or hepatic insufficiency.
* Allergy to any of the drugs used in the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Onset of sensory analgesia | 24 hours
  will be assessed by pin prick and cold application from the start of epidural infusion till scoring 1 at the 3 point scale. Assessment will be done every 5 minutes until the onset of sensory block using a 3-point scale: 0=normal sensation, 1=loss of sensation of pin prick (analgesia), and 2=loss of sensation of touch (anesthesia).
Duration of analgesia | 24 hours
  time from starting epidural infusion to the time of the first request for additional pain medication

SECONDARY OUTCOMES:
Postoperative pain score | 24 hours
  for 24 hours using the Visual Analogue Scale ranging from 0 to 10 (0 - no pain, 10 - worst pain ever) at 0, 2, 6, 12 and 24 hrs after starting epidural infusion.
Analgesic consumption | 24 hours
  during the 24 hours following epidural infusion.
The motor block | 24 hours
  will be assessed if occurred by Bromage three point score (0-3) for the lower extremity during the 24 hours following epidural infusion where 0: no motor impairment (able to move the hip, knee, and ankle joints);
  1. unable to raise either extended leg (able to move joints of knee and ankle);
  2. unable to raise extended leg and flex knee (able to move joint of ankle); 3; unable to move knee and foot.
Post operative Mean arterial Blood pressure | 24 hours
  Mean arterial pressure in mmHg will be monitored continuously and recorded just before the initiation of epidural infusion and thereafter at 2, 6, 12 and 24 hrs. postoperatively during the 24 hours following epidural infusion
Post operative Heart rate | 24 hours
  Heart rate (HR) in beats per minute (bpm) will be monitored continuously and recorded just before the initiation of epidural infusion and thereafter at 2, 6, 12 and 24 hrs. postoperatively during the 24 hours following epidural infusion
Post operative Peripheral oxygen saturation | 24 hours
  Peripheral oxygen saturation in blood (SpO2) will be monitored continuously and recorded just before the initiation of epidural infusion and thereafter at 2, 6, 12 and 24 hrs. postoperatively during the 24 hours following epidural infusion
Anticipated adverse events | 24 hours
  like postoperative nausea and vomiting during the 24 hours from the start of epidural analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Eldin E Hassan, Professor, Study Chair — Department of Anesthesia, Intensive care and pain management, Ain Shams University.; Hadeel M Abd Elhamid, Professor, Study Director — Department of Anesthesia, Intensive care and pain management, Ain Shams University.; Mohamed A Saleh, MD, Study Director — Department of Anesthesia, Intensive care and pain management, Ain Shams University.; Ibrahim A Ibrahim, MD, Study Director — Department of Anesthesia, Intensive care and pain management, Ain Shams University.
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grewal A. Dexmedetomidine: New avenues. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):297-302. doi: 10.4103/0970-9185.83670. No abstract available. PMID 21897496
- [Background] Hetta DF, Fares KM, Abedalmohsen AM, Abdel-Wahab AH, Elfadl GMA, Ali WN. Epidural dexmedetomidine infusion for perioperative analgesia in patients undergoing abdominal cancer surgery: randomized trial. J Pain Res. 2018 Oct 30;11:2675-2685. doi: 10.2147/JPR.S163975. eCollection 2018. PMID 30464585
- [Background] Kiran S, Jinjil K, Tandon U, Kar S. Evaluation of dexmedetomidine and fentanyl as additives to ropivacaine for epidural anesthesia and postoperative analgesia. J Anaesthesiol Clin Pharmacol. 2018 Jan-Mar;34(1):41-45. doi: 10.4103/joacp.JOACP_205_16. PMID 29643621
- [Background] Mohamad MF, Mohammad MA, Hetta DF, Ahmed EH, Obiedallah AA, Elzohry AAM. Thoracic epidural analgesia reduces myocardial injury in ischemic patients undergoing major abdominal cancer surgery. J Pain Res. 2017 Apr 12;10:887-895. doi: 10.2147/JPR.S122918. eCollection 2017. PMID 28442930
- [Background] Yousef AA, Salem HA, Moustafa MZ. Effect of mini-dose epidural dexmedetomidine in elective cesarean section using combined spinal-epidural anesthesia: a randomized double-blinded controlled study. J Anesth. 2015 Oct;29(5):708-14. doi: 10.1007/s00540-015-2027-7. Epub 2015 May 26. PMID 26006222
- [Background] Zhao Y, Xin Y, Liu Y, Yi X, Liu Y. Effect of Epidural Dexmedetomidine Combined With Ropivacaine in Labor Analgesia: A Randomized Double-Blinded Controlled Study. Clin J Pain. 2017 Apr;33(4):319-324. doi: 10.1097/AJP.0000000000000411. PMID 27513640
- [Background] Soliman, Rabie & Eltaweel, Moataz. (2016). Comparative study of dexmedetomidine and fentanyl as an adjuvant to epidural bupivacaine for postoperative pain relief in adult patients undergoing total knee replacement: a randomized study. Journal of Anesthesiology and Clinical Science. 5. 1. 10.7243/2049-9752-5-1.
- See also: National institute for health and clinical excellence — http://www.nice.org.uk.